CLINICAL TRIAL: NCT00839449
Title: Eicosapentaenoic Acid Cerebral Vasospasm Therapy Study (EVAS): Effect of Eicosapentaenoic Acid on Cerebral Vasospasm Following Subarachnoid Hemorrhage
Brief Title: Eicosapentaenoic Acid Cerebral Vasospasm Therapy Study
Acronym: EVAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yamaguchi University Hospital (Other)
Collaborators: Nakamura Memorial Hospital (Other); Iwate Medical University (Other); Tohoku University (Other); Ootemachi Hospital (Unknown)
Responsible Party: Eicosapentaenoic acid Cerebral Vasospasm Therapy Study (EVAS) Group, Yamaguchi University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Y-2004
Record Dates: First submitted 2009-02-04; First posted 2009-02-09 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Subarachnoid Hemorrhage; Cerebral Vasospasm
Keywords: subarachnoid hemorrhage; cerebral vasospasm; eicosapentaenoic acid
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Patients in the group A are orally administered eicosapentaenoic acid ethyl ester.
  Interventions: Drug: Eicosapentaenoic acid ethyl ester
- B (No Intervention): Patients in the group B (control) are not administered eicosapentaenoic acid ethyl ester.

INTERVENTIONS:
Drug: Eicosapentaenoic acid ethyl ester — Orally administered 900 mg eicosapentaenoic acid ethyl ester three times a day (2700 mg ⁄ day) from the surgery next day to 30 days after the onset of SAH.
  Other Names: EPADEL S900 TM (EPA ethyl ester, purity >98%)
  Arms: A

SUMMARY:
Cerebral vasospasm following subarachnoid hemorrhage (SAH) is the most common cause of morbidity and mortality. Recent studies indicate that Rho-kinase play an important role in the occurrence of such cerebral vasospasm. Eicosapentaenoic acid (EPA) inhibits sphingosylphosphorylcholine (SPC)-induced Rho-kinase activation in vitro. So this study examines whether EPA prevents cerebral vasospasm occurrence after SAH in patients.

DETAILED DESCRIPTION:
Cerebral vasospasm occasionally seen after subarachnoid hemorrhage (SAH) due to a ruptured intracranial aneurysm is the most common cause of morbidity and mortality in these cases. Recent studies indicate that Rho-kinase plays an important role in such cerebral vasospasm and that numerous agents, such as thromboxane A2 (TXA2), sphingosylphosphorylcholine (SPC) and arachidonic acid (AA), can activate Rho-kinase directly or through receptors in the cell membrane; among these agents, SPC has been described as a novel messenger for Rho-kinase-mediated Ca2+ sensitization of vascular smooth muscle contraction. Eicosapentaenoic acid (EPA) has recently been reported to inhibit SPC-induced Rho-kinase activation in vitro, and thereby vascular smooth muscle contraction, through the inhibition of Src family protein tyrosine kinases translocation. Moreover, the concentration of AA increases in the cerebrospinal fluid of patients with SAH, suggesting that this substance has a potential role in the occurrence of cerebral vasospasm following SAH, while EPA is known to change the constitution ratios of AA and EPA in cell membrane phospholipid, resulting in the inhibition of TXA2 synthesis. These observations lead us to hypothesize that EPA may inhibit cerebral vasospasm following SAH through the inhibition of Rho-kinase activation.

ELIGIBILITY:
Inclusion Criteria:

* Subarachnoid hemorrhage (SAH)
* The ruptured cerebral aneurysms conformed by cerebral angiography
* The patients with treated by craniotomy and clip application within 72h after the onset of SAH

Exclusion Criteria:

* Traumatic or mycotic aneurysms
* A history or complication of serious stroke
* Moya Moya disease
* A history of SAH
* Complication of serious heart or hepatic disease or infection or renal failure
* Malignant tumor
* Patients judged to be inappropriate by physician in charge

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-12; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cerebral vasospasms: Symptomatic vasospasm defined as documented arterial vasospasm consistent with new neurological deterioration. New low-density areas on CT scans associated with vasospasm. | Between 4 and 30 days after the onset of SAH

SECONDARY OUTCOMES:
Patient's Glasgow Outcome Scale (GOS). | At 1 month after onset of SAH.

CONTACTS AND LOCATIONS:
Overall Officials: Michiyasu Suzuki, MD, PhD, Principal Investigator — Yamaguchi University Hospital
Locations (5):
- Japan (5):
  - Ootemachi Hospital, Kitakyushu, Fukuoka
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - Iwate Medical University, Morioka, Iwate
  - Tohoku University, Sendai, Miyagi
  - Yamaguchi University Hospital, Ube, Yamaguchi

REFERENCES:
- [Derived] Yoneda H, Shirao S, Nakagawara J, Ogasawara K, Tominaga T, Suzuki M. A prospective, multicenter, randomized study of the efficacy of eicosapentaenoic acid for cerebral vasospasm: the EVAS study. World Neurosurg. 2014 Feb;81(2):309-15. doi: 10.1016/j.wneu.2012.09.020. Epub 2012 Sep 29. PMID 23032083